CLINICAL TRIAL: NCT01103739
Title: A Phase 1, Open Label, Fixed Sequence Study To Investigate The Effect Of Multiple Doses Of PF-04531083 On Simvastatin And Simvastatin Acid Pharmacokinetics Following Single Dose Of Simvastatin in Healthy Volunteers
Brief Title: To Explore The Potential For PF-04531083 To Effect The Blood Concentrations Of Simvastatin And Its Main Acid Metabolite Following Co-Administration Of Both Medications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B1351007
Record Dates: First submitted 2010-02-26; First posted 2010-04-15 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Pain
Keywords: pharmacokinetics; drug-drug interaction
MeSH Terms: conditions — Chronic Pain | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cohort 1 (Experimental)
  Interventions: Drug: PF-04531083; Drug: simvastatin
- cohort 2 (Experimental)
  Interventions: Drug: PF-04531083; Drug: simvastatin

INTERVENTIONS:
Drug: PF-04531083 — PF-04531083: 100mg to be dosed twice daily as a suspension from Day 2 through Day 14 of the study.
  Arms: cohort 1
Drug: simvastatin — Simvastatin: a single 20mg tablet to be given on Days 1 and 14 of the study.
  Arms: cohort 1
Drug: PF-04531083 — PF-04531083: a dose to be selected depending on results from Cohort 1 to be dosed twice daily as a suspension from Day 2 through Day 14 of the study.
  Arms: cohort 2
Drug: simvastatin — Simvastatin: a single 20mg tablet to be given on Days 1 and 14 of the study.
  Arms: cohort 2

SUMMARY:
The purpose of this study is to quantify the effect of multiple doses of PF-04531083 on the pharmacokinetics (PK) of co-administered single dose simvastatin.

DETAILED DESCRIPTION:
observational- quantify any effects of PF_04531083 on the PK of Simvastatin

ELIGIBILITY:
Inclusion Criteria:

* young
* healthy
* male and female volunteers

Exclusion Criteria:

* Elderly
* Patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of simvastatin. AUC, Cmax and half life. | days 1 and 14 of study
Pharmacokinetics of simvastatin acid. AUC, Cmax and half life. | days 1 and 14 of study
Trough concentrations of PF-04531083 2, 4, 7, 11 and 14 days post commencement of dosing | days 2, 4, 7, 11 and 14 of the study

SECONDARY OUTCOMES:
safety and tolerability of PF-04531083 and simvastatin. Vital signs, laboratory tests and adverse events | days 1 and 15 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351007&StudyName=To%20Explore%20The%20Potential%20For%20PF-04531083%20To%20Effect%20The%20Blood%20Concentrations%20Of%20Simvastatin%20And%20Its%20Main%20Acid%20Metabolite%20Following%20Co-Adm